CLINICAL TRIAL: NCT06514664
Title: Evaluation of the Effects of Probiotic Toothpastes on Periodontal Health
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc.Prof.Dr., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-03/08
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Diseases; Periodontitis; Gingivitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Use of probiotic toothpaste + smoking patient
  Interventions: Other: Using Probiotic Toothpaste
- Group 2 (No Intervention): Use of regular toothpaste + smoking patient
- Group 3 (Experimental): Use of probiotic toothpaste + non-smoking patient
  Interventions: Other: Using Probiotic Toothpaste
- Group 4 (No Intervention): Use of regular toothpaste + non-smoking patient

INTERVENTIONS:
Other: Using Probiotic Toothpaste — Scaling and root planing (Phase 1 = non-surgical periodontal treatment) are performed in all patient groups.
  Depending on the study groups, regular or probiotic toothpaste will be used. Toothpaste is instructed to be used twice a day
  Arms: Group 1; Group 3

SUMMARY:
This controlled, randomized clinical study aims to evaluate the possible effects of probiotic toothpaste on the success of periodontal treatment in smokers and non-smokers with clinical data.

The main question(s) it aims to answer are:

Does applying probiotic toothpaste in addition to periodontal treatment have a positive effect on the gingival of periodontitis patients who are smokers and non-smokers?

The study includes four groups; Group 1: Use of probiotic toothpaste + smoking patient Group 2: Use of regular toothpaste + smoking patient Group 3: Use of probiotic toothpaste + non-smoking patient Group 4: Use of regular toothpaste + non-smoking patient

DETAILED DESCRIPTION:
Periodontitis is characterized by the progressive destruction of all periodontium structures that support the teeth, including periodontal connective tissue and alveolar bone, caused by dental biofilm, resulting in irreversible damage. Severe periodontitis has become a public health problem that affects approximately 11% of the world's population, that is, 743 million people. When left untreated, it reduces the quality of life and leads to tooth loss. In addition to being a common cause of tooth loss, severe periodontitis has been reported to be a predisposing factor in the development of major systemic diseases such as atherosclerosis, cerebrovascular disease, diabetes, rheumatoid arthritis, Alzheimer's disease and some cancers, and increases the risk of adverse pregnancies (low birth weight, preterm birth). Periodontal inflammation is caused by the presence of gram-negative anaerobic bacteria called "red complex" in the subgingival plaque. Red complex bacteria include Porphyromonas gingivalis, Tannerella forsythia and Treponema denticola, which are responsible for the onset and development of periodontal disease and are found predominantly in the deep periodontal pockets of patients with periodontitis.

In addition, genetic and environmental factors may increase an individual's susceptibility to periodontal disease. The patient's smoking and diabetes mellitus are risk factors for periodontitis. Smoking is the most important environmental risk factor for periodontitis. When subgingival biofilms of nonsmokers/former smokers were compared with smokers, smokers exhibited a higher prevalence of red complex bacteria. Additionally, it has been reported that the potential negative effect of smoking on immune cells, especially neutrophils, makes the individual more susceptible to periodontitis. It has been observed that periodontitis patients who smoke have more alveolar bone and attachment loss than non-smokers. The main goal of periodontal treatment in patients diagnosed with periodontitis is based on removing subgingival biofilm and dental calculus. Before applying surgical periodontal treatment, which is the second step, the first step is non-surgical periodontal treatment and is a prerequisite for deciding to proceed to the surgical stage. In addition to non-surgical periodontal treatment, Local and/or systemic antibiotics, anti-inflammatory drugs, photodynamic therapy, laser, probiotics, prebiotics and synbiotics, statins, ozone therapy, epigenetic therapy, and omega 3-6 can be used. Probiotics modulate the oral microbiota by integrating beneficial bacteria into oral biofilms and preventing the treatment of oral microbial diseases. Probiotics are defined as live microorganisms that provide health benefits when administered in sufficient amounts. The most common probiotic bacteria are Lactobacillus and Bifidobacterium species. Probiotic bifidobacteria have antimicrobial activity against periodontal pathogenic bacteria P. gingivalis and Fusobacterium nucleatum. In an in vitro study by Jasberg et al., it was shown that species belonging to the genus Bifidobacterium could strongly adhere to the subgingival biofilm and significantly reduce the number of Porphyromonas gingivalis. All bifidobacteria integrated well into subgingival biofilms consisting of Porphyromonas gingivalis, Actinomyces naeslundii, and Fusobacterium nucleatum, but only significantly reduced the number of P.gingivalis in biofilms. In the systematic review and meta-analysis evaluating the additional use of probiotics in patients with chronic periodontitis, seven clinical studies evaluating the effectiveness of probiotics as an aid in scaling and root planing were included. While four studies showed additional benefits of probiotics in reducing pocket depth and providing clinical attachment gain, Three studies showed no significant differences. In addition, the difference between the average clinical attachment gain of the patients during the long-term follow-up phases was found to be significant. Today, studies show that probiotic toothpaste effectively prevents infectious diseases such as caries or periodontal disease. However, there are no studies on the effect of smoking on the effectiveness of toothpaste.

Probiotic Toothpaste Content: Glycerin, Hydrated Silica, Aqua, Aloe Barbedensiz, Leaf Juice, Citric Acid, Potassium Sorbate, Sodium Benzoate, Xanthan Gum, B.Coagulans BC4, Xylitol, Sodium Coco-Sulfate, Sodium Hydroxide, Lavandula AngusTifolia (Lavender) Contains Oil (Linalool).

OHIP-14 survey: The effect of the treatment on the patient's quality of life is evaluated with a 14-question survey asked before and one month after non-surgical periodontal treatment.

Periodontal indexes will be taken from all patients in the study group after taking systemic and dental anamnesis. At the first examination session, study samples will be taken, clinical periodontal measurements (plaque index, gingival index, bleeding index, pocket depth, attachment loss, were used to evaluate the periodontal status in 6 regions of each tooth (mesio-buccal, buccal, disto-buccal, disto-palatal, palatal, mesio-palatal) with the Williams periodontal probe (Hu-Friedy, USA) will be measured and recorded) and the oral health effective profile-14 (OHIP-14) questionnaire will be recorded. Afterward, all teeth will be cleaned with an ultrasonic device, and oral hygiene training will be given to the patients. Patients will be taught how to brush their teeth using the modified Bass technique and how to use an interdental brush. In the second session, tooth brushing and interdental brush usage will be checked, and if sufficient, dental floss training will be given; if inadequate, brush usage will be explained again.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years old
2. Pocket depth ≥ 4 mm and clinical attachment loss ≥ 1 mm in at least 5 teeth, bleeding score on probing 20%, and widespread bone loss that can be diagnosed radiographically.
3. Absence of any systemic disease
4. Having at least 14 natural teeth
5. Diagnosing periodontitis as a result of clinical and radiological examinations
6. Volunteering to participate in the research and signing the consent form prepared in accordance with the Declaration of Helsinki.

Exclusion Criteria:

1. Being outside the specified age range
2. Being pregnant or lactating
3. Having used antibiotics for any reason in the last 3 months
4. Having had periodontal treatment in the last 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Periodontal pocket depth changes | 3 month follow up
  Periodontal pocket depth changes will be measured with periodontal probe at baseline and third month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Guler Ayyildiz, Principal Investigator — Kutahya Health Science University; Ahu Uraz Corekci, Principal Investigator — Izmir Democracy University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If contacted, the principal researcher's evaluation will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Six months after the study is completed and published
Access Criteria: If contacted, the principal researcher's evaluation will be shared.